CLINICAL TRIAL: NCT04131790
Title: Improving Social Connectedness in Home Delivered Meals Clients
Brief Title: Tele-BA for Home-Delivered Meals Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Martha L. Bruce, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D19169
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Social Isolation
Keywords: Loneliness; Homebound; Behavioral Activation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Behavioral Activation (Experimental): Manualized Behavioral Activation (BA) protocol delivered via videoconferencing by a trained BA interventionist; 5 sessions over 5 weeks, up to 1-hour in length. The interventionist guides participants in learning BA skills, focusing on strategies to decrease barriers to social connectedness (e.g., limited mobility, inadequate caregiving resources).
  Interventions: Behavioral: Tele-Behavioral Activation
- Tele-Friendly Visiting (Active Comparator): Friendly Visitor (FV) calls delivered via videoconferencing by a trained FV interventionist; 5 sessions over 5 weeks, up to 1-hour in length. The interventionist provides social support to participants through good listening and provision of genuine regard.
  Interventions: Behavioral: Tele-Friendly Visiting

INTERVENTIONS:
Behavioral: Tele-Behavioral Activation — Five 1-hour sessions of BA delivered by a trained interventionist via video-conferencing
  Arms: Tele-Behavioral Activation
Behavioral: Tele-Friendly Visiting — Five 1-hour FV sessions delivered by a trained interventionist via video-conferencing
  Arms: Tele-Friendly Visiting

SUMMARY:
The purpose of this study to evaluate aging-service integrated, video-conference-based approaches to improve homebound seniors' social engagement and activities.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Clients of the Meals on Weals program
* ≥60 years old
* Score between 6-9 on the Hughes three-item version of the UCLA Loneliness Scale

Exclusion Criteria:

* Dementia, as indicated by a score > 3 on the Six Item Screen
* Clinically significant depression, as indicated by a score ≥15 on the Patient Health Questionnaire (PHQ-9)
* Active suicide risk, as indicated by a positive response on any item of the Columbia Suicide Severity Rating Scale (C-SSRS)
* Uncorrectable hearing or vision impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change over time in social support measured using the Duke Social Support Index (DSSI) | Baseline, 6-week follow-up (immediately post-intervention), 12-week follow up (12 weeks post-intervention), 12-month follow-up (12-months post-intervention).
  A 10-item self-report questionnaire used to measure an individual's satisfaction with social support using a Likert scale (3-point scale, where anchor labels are specified for each item). This scale consists of two subscales: 4-item social interaction (objective support) scale and 6-item satisfaction with social support (subjective support) subscale. Total scores are calculated by summing responses to items across all items; total scores range 10-30.
Change over time in perceived social isolation measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Social Isolation Scale | Baseline, 6-week follow-up (immediately post-intervention), 12-week follow up (12 weeks post-intervention), 12-month follow-up (12-months post-intervention).
  An 8-item self-report questionnaire used to measure perceived social isolation using a Likert scale (5-point scale: 'never' = 1 to 'always' = 5). Total raw scores range from 8-40; raw scores are converted to T-scores using an appendix (T-scores are standardized scores that have a mean of 50 and SD of 10). Higher T-score values represent greater perceived social isolation.

SECONDARY OUTCOMES:
Change over time in depression symptomatology measured using the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 6-week follow-up (immediately post-intervention), 12-week follow up (12 weeks post-intervention), 12-month follow-up (12-months post-intervention).
  A 9-item self-report questionnaire used to measure symptoms of depression. Items are rated using a Likert scale (4-point scale: 'not at all' = 0 to 'nearly every day' = 3). Total scores are calculated by summing responses to items 1-9; total scores range 0-27.
Change over time in functional disability measured using the World Health Organization Disability Assessment Schedule (WHODAS 2.0) | Baseline, 6-week follow-up (immediately post-intervention), 12-week follow up (12 weeks post-intervention), 12-month follow-up (12-months post-intervention).
  A 12-item self-report questionnaire used to assess functioning in six domains of life:
  Domain 1: Cognition - understanding and communicating Domain 2: Mobility - moving and getting around Domain 3: Self-care - attending to one's hygiene, dressing, eating and staying alone Domain 4: Getting along - interacting with other people Domain 5: Life activities - domestic responsibilities, leisure, work and school Domain 6: Participation - joining in community activities, participating in society.
  Items are rated using a Likert scale (5-point scale: 'none' = 0 to 'Extreme/cannot do' = 4). Total scores are calculated by summing responses to items 1-12; total scores range 0-48.

OTHER OUTCOMES:
Acceptance of the Tele-BA intervention using a modified version of the Treatment Evaluation Inventory (TEI) | 6-weeks follow-up (immediately post-intervention)
  An 11-item self-report questionnaire used to measure intervention acceptability. For this project, reference to "Treatment" will be substituted with "Tele-BA." Items are rated using a 7-point Likert scale. Response values range 1-7 with different verbal anchors for each item. Total scores are calculated by summing responses to items 1-11; total scores range 11-77. The TEI consists of an 8-item General Acceptability subscale and a 3-item Negative Aspects (e.g., discomfort) subscale.
Change over time in social activities participation using the Social Engagement/Activities Questionnaire (SEAQ) | Baseline, 6-week follow-up (immediately post-intervention), 12-week follow up (12 weeks post-intervention), 12-month follow-up (12-months post-intervention).
  A 10-item self-report questionnaire used to measure homebound older adults' participation in a range of social-group activities, interpersonal interaction activities with family and friends, and solitary activities while taking account of their physical and functional health limitations and social circumstances under which they live. Items are rated using a Likert scale (6-point scale: 'not at all' = 0 to 'every day' = 5). Total scores are calculated by summing responses to items 1-10; total scores range 0-50.
Change over time in coping strategies using the Brief COPE | Baseline, 6-week follow-up (immediately post-intervention), 12-week follow up (12 weeks post-intervention), 12-month follow-up (12-months post-intervention).
  A 16-item self-report questionnaire used to measure use of coping strategies for difficult situations. Items are rated using a Likert scale (4-point scale: 'not at all' = 0 to 'a lot' = 3). Total scores are calculated by summing responses to items 1-16; total scores range 0-48.

CONTACTS AND LOCATIONS:
Overall Officials: Martha L Bruce, PhD, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
At this time there are no plans to share individual patient data.

REFERENCES:
- [Derived] Choi NG, Pepin R, Marti CN, Stevens CJ, Bruce ML. Improving Social Connectedness for Homebound Older Adults: Randomized Controlled Trial of Tele-Delivered Behavioral Activation Versus Tele-Delivered Friendly Visits. Am J Geriatr Psychiatry. 2020 Jul;28(7):698-708. doi: 10.1016/j.jagp.2020.02.008. Epub 2020 Mar 2. PMID 32238297